CLINICAL TRIAL: NCT01917422
Title: Clinical Specimens Testing Program of Dengue Antigen Detection Reagents
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-2012-03-14(II)
Record Dates: First submitted 2012-09-28; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — no biospecimens are to be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
Dengue virus serological reagent, included antigen and antiserum, is a serum test for identification of serum antibodies to dengue virus.

DETAILED DESCRIPTION:
The developed assay helps to diagnose diseases caused by this virus and to provide information on disease epidemiology. This virus is mainly transmitted by mosquito bites to people and will make flu-like symptoms, including fever, fatigue, cough and headache, which can cause severe hemorrhagic dengue.

ELIGIBILITY:
Inclusion Criteria:A total of 95 cases and 100 controls (suspected cases(>50 %) and normal subjects) are expected to enroll.

1. Case group: adults having a medical visit or admission due to dengue / dengue hemorrhagic fever / dengue shock syndrome, and medical care of by (defined by CDC). Any of the following positive test results for the case of 100 adults.

   1. clinical specimens (blood) isolated and identified dengue virus.
   2. clinical specimens positive for molecular detection of nucleic acids.
   3. serological antigen (referring to non-structural proteins of dengue virus non-structural protein 1, NS1) testing positive (based on the test of Bio-Rad DENGUE NS1 Ag STRIP).
   4. paired serum (restored period and acute phase), the dengue virus specific immunoglobulin M or immunoglobulin G antibodies or negative or ≧ 4 times increase.
2. Suspected cases: adults having medical visits or admissions due to infectious disease, but their NS1 (based on the test of Bio-Rad DENGUE NS1 Ag STRIP), immunoglobulin G,immunoglobulin M, real time-Polymerase chain reaction testing were negative.
3. Control group: adults without having medical visits or admissions due to Fever. - Exclusion Criteria:non-adult case -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The samples are obtained from the Kaohsiung Medical University Chung-Ho Memorial Hospital in Kaohsiung, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical specimens testing program of dengue antigen detection reagents | one year
  Calculate two products of the dengue immune detection accuracy, sensitivity, specificity, false positive, false negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshiung, Taiwan